CLINICAL TRIAL: NCT04998799
Title: Current Practices on Antithrombotic Therapy in Hospitalised and Discharged Patients With COVID-19
Brief Title: Practice Variation on Antithrombotics in COVID-19
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Head Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: ATCOVIDIndia
Record Dates: First submitted 2021-08-08; First posted 2021-08-10 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pneumonia; Thrombosis; COVID-19 Acute Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome (SARS) Pneumonia
Keywords: Anticoagulation in COVID-19; Anticoagulants; SARS-CoV-2; Coronavirus Disease 2019; Management of COVID-19
MeSH Terms: conditions — Thrombosis; Severe Acute Respiratory Syndrome; Pneumonia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Current clinical practices of participating physicians — Current clinical practice of participating physicians on management of antithrombotics for COVID-19 during hospitalisation and post-discharge

SUMMARY:
Evidence suggests coronavirus disease 2019 (COVID-19) is associated with an increased incidence of thromboembolic manifestations. Various guidelines on managing antithrombotics in COVID-19 either provided conflicting guidance or unclear recommendations for post-discharge thromboprophylaxis.

The investigators aim to collect the current practices in India among physicians on antithrombotic therapy for hospitalised patients with COVID-19 and after discharge from the hospital.

DETAILED DESCRIPTION:
Immune dysregulation plays a crucial role in the development of severe coronavirus disease 2019 (COVID-19). The autopsy of lungs in deceased COVID-19 patients showed micro thrombosis and inflammatory infiltrates similar to acute respiratory distress syndrome (ARDS). Reports of increased incidence of arterial or venous thrombosis with COVID-19 made initial recommendations regarding using higher doses of anticoagulation. The markers of thrombosis like D-dimer, platelet count, fibrinogen are also increased in patients with COVID-19 along with other inflammatory markers. The pathophysiology of coagulopathy of COVID-19 is still under research. It is likely multi-factorial involving Inflammation, hypoxia, endothelial dysfunction, direct viral cytopathic effect, platelets and complement activation, derangement of the renin-angiotensin-aldosterone pathway.

From the inception of the pandemic, the physicians started using various antithrombotic with higher than prophylactic doses to treat the prothrombotic state. In the absence of clear guidance with conflicting evidence, there is considerable variation in the practices of physicians managing COVID-19.

The investigators are planning for a nationwide multicentre cross-sectional survey on understanding participating physicians practices on the choice of different antithrombotics available in India as of August 2021.

The survey will have three sections: 1. Demographics 2. Antithrombotics in hospitalised patients 3. Antithrombotics after discharge from the hospital

The investigators intend to involve 1000 physicians from different specialities with the help of the steering committee.

ELIGIBILITY:
Inclusion Criteria:

• Physicians involved in the management of adult hospitalised patients with COVID-19 in India

Exclusion Criteria:

* Pediatricians
* Physicians involved in the out-patient management of COVID-19
* Refused to participate

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians from different specialities like Internal Medicine, Pulmonary Medicine, Anesthesiologists, Critical Care Medicine will be recruited through snowballing sampling. A web-based cross-sectional survey will be circulated among the target population by the investigators through e-mail and social media channels.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Choice, dose, and indication of antithrombotics for management of COVID-19. | two weeks
  Through web-based cross-sectional survey will capture the practices of physicians on choice, dose, and indication of antithrombotics for management of COVID-19 during hospitalisation and post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Nasa, MD EDICM, Principal Investigator — NMC Specialty Hospital, Dubai, UAE
Locations (1):
- Reliance Hospital, Mumbai, Mumbai, Mahrastra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandra A, Chakraborty U, Ghosh S, Dasgupta S. Anticoagulation in COVID-19: current concepts and controversies. Postgrad Med J. 2022 May;98(1159):395-402. doi: 10.1136/postgradmedj-2021-139923. Epub 2021 Apr 13. PMID 33850011
- [Background] Fontelo P, Bastola MM, Zheng Z, Baik SH. A review of thromboembolic events in hospitalized COVID-19 patients. Thromb J. 2021 Jun 29;19(1):47. doi: 10.1186/s12959-021-00298-3. PMID 34187490
- [Background] Jagiasi B, Nasa P, Chanchalani G, Ahmed A, Ak AK, Sodhi K, Mangal K, Singh MK, Gupta N, Bidkar PU, Tyagi RS, Khanikar RG, Tripathy S, Khanzode S, Subba Reddy K, Saigal S, Sivakumar VA, Javeri Y, Tekwani SS. Variation in therapeutic strategies for the management of severe COVID-19 in India: A nationwide cross-sectional survey. Int J Clin Pract. 2021 Oct;75(10):e14574. doi: 10.1111/ijcp.14574. Epub 2021 Jul 18. PMID 34171154
- [Background] Liu Y, Cai J, Wang C, Jin J, Qu L. A systematic review and meta-analysis of incidence, prognosis, and laboratory indicators of venous thromboembolism in hospitalized patients with coronavirus disease 2019. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1099-1111.e6. doi: 10.1016/j.jvsv.2021.01.012. Epub 2021 Jan 30. PMID 33529719